CLINICAL TRIAL: NCT01051154
Title: The Effect of Enteral Administration of Polyunsaturated Omega-3 Fatty Acids on Nutritional Status; the Treatment Toxicity and Early Mortality in Children With Acute Lymphoblastic Leukemia - a Controlled Study
Brief Title: Effect of Enteral Docosahexaenoic Acid Administration in Children With Acute Lymphoblastic Leukemia
Acronym: DHA-ALL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Collaborators: National Council of Science and Technology, Mexico (Other); Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, María de Lourdes Barbosa Cortés, Associated Researcher, Coordinación de Investigación en Salud, Mexico
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009-785-107; 113742 (Other Grant/Funding Number: CONACyT)
Record Dates: First submitted 2010-01-15; First posted 2010-01-18 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-08

CONDITIONS: Acute Lymphoblastic Leukemia; Malnutrition
Keywords: Docosahexaenoic acid; Nutritional status; Acute lymphoblastic leukemia; Long chain polyunsaturated fatty acids; n-3 fatty acids; Remission-induction phase
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Malnutrition | interventions — Docosahexaenoic Acids; Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Docosahexaenoic acid (DHA) (Active Comparator): This group will be receive the DHA supplement
  Interventions: Dietary Supplement: Docosahexaenoic acid (DHA)
- Placebo (Placebo Comparator): This group will be receive placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Docosahexaenoic acid (DHA) — Children will be received either fish oil capsules (DHA group) or placebo capsules (placebo group) which is visually indistinguishable from DHA capsules (softgel). Each child will be receiving 100 mg/kg/day or placebo capsules without docosahexaenoic acid, during the first three months of treatment.
  Other Names: omega 3 fatty acids; n-3 LC-PUFAs; long chain polyunsaturated fatty acids
  Arms: Docosahexaenoic acid (DHA)
Dietary Supplement: Placebo — Children will be received either fish oil capsules (DHA group) or placebo capsules (placebo group) which is visually indistinguishable from DHA capsules (softgel). Each child will be receiving 100 mg/kg/day or placebo capsules without docosahexaenoic acid, during the first three months of treatment.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate if enteral docosahexaenoic acid (DHA) administration during the first three months of treatment reduces the deterioration of nutritional status, treatment toxicity and early mortality in children with acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
Cancer is often associated with malnutrition.The most of children with cancer loss weight, and 50-80% of patients with cancer experience morbidity and mortality as a result of progressive wasting.

As a consequence of malnutrition, patients with cancer may have a poorer outcome, reduced effectiveness of chemotherapy and increased risk of chemotherapy-induced toxicity compared to those who are well nourished at diagnosis. On the other hand, in the recent years, there has been increased focus on the role of long chain polyunsaturated fatty acids and their effect on prevention and treatment of several diseases. The results of animal studies and adults with cancer have demonstrated that the consumption of long chain polyunsaturated fatty acids can slow the growth of cancer, increase the efficacy of chemotherapy and reduce loss weight and the side effects of the chemotherapy.

Beneficial effects of enteral long chain polyunsaturated fatty acids has been reported in adults with cancer. However, in children with cancer the scientific reports are scarce; therefore, is necessary to evaluate if the long chain polyunsaturated fatty acids administration in children with acute lymphoblastic leukemia has the same effects on clinical and nutritional outcomes that have been previously showed by different studies in adults with cancer.

ELIGIBILITY:
Inclusion Criteria:

* Children with acute lymphoblastic leukemia diagnosis
* Authorization from both parents or legal guardian for recruiting of the child into the study with consent signed form after the purpose and procedures have been explained
* Must be able to swallow capsules of DHA or placebo
* Malnutrition

Exclusion Criteria:

* Patients had received radiotherapy or chemotherapy
* Parents who decide to decline of the study

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2010-09; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Nutritional status will be determined by the register of anthropometrical measurements, body composition by DEXA, and biochemical markers. | At the time of diagnosis and the first three months of treatment

SECONDARY OUTCOMES:
Treatment toxicity measured by complications and haematological and biochemical outcomes,will be evaluated according to criteria established by the World Health Organization. | The first three months of treatment
Early mortality will be considered as the difference between the total number of individuals alive at the end of follow-up (3 months) unless the initial number of patients included in the study for each group | The first three months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Maria de Lourdes Barbosa-Cortes, MSc, Principal Investigator — Instituto Mexicano del Seguro Social
Locations (1):
- Unit of Research in Nutrition, Pediatric Hospital, Instituto Mexicano del Seguro Social, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Larsson SC, Kumlin M, Ingelman-Sundberg M, Wolk A. Dietary long-chain n-3 fatty acids for the prevention of cancer: a review of potential mechanisms. Am J Clin Nutr. 2004 Jun;79(6):935-45. doi: 10.1093/ajcn/79.6.935. PMID 15159222
- [Derived] Barbosa-Cortes L, Martinez-Vieyra X, Mejia-Arangure JM, Lopez-Alarcon M, Martin-Trejo J, Delgadillo-Portillo S, Guzman-Castro B, Delgadillo-Portillo J, Atilano-Miguel S, Rodriguez-Cruz M, Maldonado-Hernandez J, Anoveros-Barrera A, Solis-Labastida KA, Espinoza-Hernandez L, Nunez-Villegas NN, Jimenez-Hernandez E, Bautista-Martinez BA, Juarez-Moya A, Hernandez-Pinon Z, Perez-Casillas RX. Pilot study on the effect of supplementation with long-chain omega-3 polyunsaturated fatty acids on body composition in children with acute lymphoblastic leukemia: randomized clinical trial. Clin Nutr. 2023 Sep;42(9):1759-1769. doi: 10.1016/j.clnu.2023.06.022. Epub 2023 Jul 13. PMID 37549598
- [Derived] Barbosa-Cortes L, Atilano-Miguel S, Martin-Trejo JA, Jimenez-Aguayo E, Martinez-Becerril FI, Lopez-Alarcon M, Mejia Arangure JM, Maldonado-Hernandez J, Delgadillo-Portillo S, Guzman-Castro B, Delgadillo-Portillo J, Anoveros-Barrera A, Solis-Labastida KA, Bautista-Martinez BA, Juarez-Moya A, Hernandez-Pinon Z, Espinoza Hernandez LE, Nunez-Villegas NN, Jimenez-Hernandez E, Perez-Casillas RX. Effect of long-chain omega-3 polyunsaturated fatty acids on cardiometabolic factors in children with acute lymphoblastic leukemia undergoing treatment: a secondary analysis of a randomized controlled trial. Front Endocrinol (Lausanne). 2023 Apr 14;14:1120364. doi: 10.3389/fendo.2023.1120364. eCollection 2023. PMID 37124732